CLINICAL TRIAL: NCT01481298
Title: Value of Different Myocardial Parameters to Differentiate Left Ventricular Noncompaction Cardiomyopathy From Other Cardiomyopathies and Healthy Controls by Cardiac Magnetic Resonance
Brief Title: Value of Cardiac Magnetic Resonance (CMR) Derived Parameters for Diagnosing Left Ventricular Non-compaction Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Matthias Grothoff, M.D., Dr. med., University of Leipzig
Other Study IDs: LVNC 2011
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Left Ventricular Non-compaction Cardiomyopathy; Left Ventricular Failure; Left Ventricular Hypertrophy
MeSH Terms: conditions — Heart Failure; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- LVNC: 12 patients with left ventricular non-compaction cardiomyopathy
- HCM: 10 patients with hypertrophic cardiomyopathy
- DCM: 11 patients with dilatative cardiomyopathy
- controls: 24 healthy controls

SUMMARY:
Left ventricular non-compaction (LVNC) is a rare cardiomyopathy characterized by numerous excessively prominent left ventricular (LV) trabeculation and deep intertrabecular recesses communicating with the ventricular cavity and severely altering myocardial structure. Although most authors assume a developmental arrest in embryogenesis as the underlying pathology, the mechanisms of LVNC are not fully understood yet. Several gene mutations have been identified to be linked with LVNC and an autosomal dominant inheritance pattern is frequent To date the most commonly used imaging tool for diagnosing LVNC is echocardiography applying the criteria established by Jenni and coauthors However, qualitative parameters to differentiate normal compaction of the myocardium in healthy subjects from LVNC or from other cardiomyopathies like dilative cardiomyopathy (DCM) or hypertrophic cardiomyopathy (HCM) may fail due to highly variable LV trabeculation. Therefore, absolute quantification should be performed. Cardiac magnetic resonance (CMR) has been reported as a promising imaging modality to characterize patients with LVNC as it provides both a high spatial resolution and a good contrast between trabeculation and blood pool Jacquier et al. recently described a value of trabeculated LV myocardial mass above 20% of the global mass of the LV to be highly sensitive and specific for LVNC However, in their approach, a substantial degree of the LV cavity was included into calculated trabecular LV mass and led to systemic overestimation of the latter. Furthermore, the role and prognostic value of myocardial scarring as assessed by delayed enhancement (DE) CMR was not evaluated.

The aim of the retrospective study was to establish revised and extended CMR criteria to distinguish LVNC from DCM, HCM and a group of healthy controls and to improve the assessment of trabeculated mass by excluding intertrabecular blood pool.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular non-compaction cardiomyopathy
* dilatative cardiomyopathy
* hypertrophic cardiomyopathy or healty controls

Exclusion Criteria:

* contraindications for magnetic resonance imaging like pacemakers or other metallic implants

Ages: 14 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Twelve patients (3 male, 27%) with proven LVNC, two with familial LVNC, were included into the study. The patients initially presented with symptoms of heart failure and were referred to the department of cardiology for further evaluation. All patients underwent echocardiography performed by experienced specialists and fulfilled the LVNC criteria of Jenni. CMR imaging was performed within 3 days after echocardiography. Exclusion criteria were co-existing cardiac anomalies and usual CMR contraindications such as implanted defibrillators/pacemakers. The investigators furthermore included 10 consecutive patients (4 male, 36%) with HCM and 11 consecutive patients (3 male, 27%) with DCM. The diagnosis of HCM and DCM was established according to current guidelines Patient parameters were compared to a control group of 25 healthy age matched volunteers (12 male, 48%) without history of cardiovascular disease and without clinical symptoms.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2004-12; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany